CLINICAL TRIAL: NCT05833178
Title: The Effect of Blood Tests Performed Within the Routine Protocol in the Surgical Intensive Care Unit on Hemoglobin Levels
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, dilan akyurt, Specialist of Anaesthesiology and Reanimasion, Samsun University
Other Study IDs: SUKAEK-2023 5/22
Record Dates: First submitted 2023-04-15; First posted 2023-04-27 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Anemia
Keywords: Intensive care unit; Routine blood sample; Overdrawn
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Drawn Blood Volume — Hemoglobine Changes

SUMMARY:
Examination of blood samples is inevitable in intensive care units. Routine blood samples can be an important cause for anemia. In this study, we aimed to examine how our blood collection routine affects hemoglobin values.

DETAILED DESCRIPTION:
Blood tests for follow-up and treatment are widely used in intensive care units (ICU). Although its etiology is very diverse, phlebotomy performed due to frequent laboratory tests is among the preventable causes of anemia. In this observational study, blood tests performed on patients treated in intensive care units followed up in our clinic between 01.April.2023 - 31.May.2023 (2 months) will be examined. Patients' age, presence of additional disease, indication for admission to the unit, Acute Physiology and Chronic Health Assessment II (APACHE II), Sequential Organ Failure Assessment (SOFA) and Glasgow coma scale (GCS), hemoglobin values will be recorded. The daily blood test will record the amount of blood drawn for analysis (in milliliters), where it was taken from (peripheral, central venous or arterial catheter), and the amount of excess blood. Statistical analysis will be performed in terms of patient characteristics, routine blood volumes and development of anemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in the intensive care unit for more than 48 hours, ≥18-year-old

Exclusion Criteria:

* Patients not followed up by our clinic,≤18-year-old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who were followed up in the intensive care unit by our clinic and treated for more than 48 hours were included in the study.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of blood volume drawn for daily routine in intensive care | 2 months
  Daily routine blood test and blood volume determination in intensive care patients

SECONDARY OUTCOMES:
Anemia | 2 months
  Evaluation of how daily routine blood drawn affects patients' hemoglobin values in intensive care patients

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa SÜREN, Study Director — Samsun University
Locations (1):
- Dilan Akyurt, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Helmer P, Hottenrott S, Steinisch A, Roder D, Schubert J, Steigerwald U, Choorapoikayil S, Meybohm P. Avoidable Blood Loss in Critical Care and Patient Blood Management: Scoping Review of Diagnostic Blood Loss. J Clin Med. 2022 Jan 10;11(2):320. doi: 10.3390/jcm11020320. PMID 35054014
- [Background] Siegal DM, Manning N, Jackson Chornenki NL, Hillis CM, Heddle NM. Devices to Reduce the Volume of Blood Taken for Laboratory Testing in ICU Patients: A Systematic Review. J Intensive Care Med. 2020 Oct;35(10):1074-1079. doi: 10.1177/0885066618810374. Epub 2018 Nov 27. PMID 30482081
- See also: Choosing Wisely — http://ccsconline.org/images/CCSC-Choosing-Wisely.pdf